CLINICAL TRIAL: NCT00694330
Title: A Phase I Study of Vaccination With Lethally Irradiated Glioma Cells Mixed With GM-K562 Cells in Patients Undergoing Craniotomy For Recurrent Tumor
Brief Title: Vaccination With Lethally Irradiated Glioma Cells Mixed With GM-K562 Cells in Patients Undergoing Craniotomy For Recurrent Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, William T. Curry, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-349
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-03

CONDITIONS: Glioma
Keywords: vaccine; GM-K562; malignant glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GM-K562 Vaccination (Experimental)
  Interventions: Biological: GM-K562 Vaccination

INTERVENTIONS:
Biological: GM-K562 Vaccination — Lethally irradiated autologous glioma cells combined with GM-K562 cells as vaccine therapy given once a week for three weeks then every other week.

SUMMARY:
This research study is testing the safety of a vaccination of cells called GM-K562 cells mixed with the participants own irradiated tumor cells. The GM-K562 cells have been modified in the laboratory to secrete the protein GM-CSF. This protein can be effective in stimulating an immune response to cancer. This newly developed vaccine may stop cancer cells from growing.

DETAILED DESCRIPTION:
* Participants will undergo a craniotomy (brain surgery) to remove as much of the tumor as possible from their brain. A pathologist will examine the tissue to determine whether the cells are viable. If not, we will not be able to make the vaccine and the participant will not be eligible to proceed with this treatment protocol.
* The dose of the vaccine will be determined by the number of tumor cells that we are able to collect from the surgery. We will also be trying to determine the appropriate number of GM-K562 cells that can be given safely. We will do this by assigning groups of participants to different dose levels of GM-K562.
* For the first three weeks of this study, vaccines will be given once each week. After the first three weeks, vaccines will be given every other week.
* Before the first and after the fourth vaccinations, a small amount of the participants own irradiated tumor cells will be injected under their skin to see if their immune system will react against it. If the participant develops a rash, they may be asked to undergo a small skin biopsy for additional evaluation. These biopsies are optional.
* During the course of the study, we will also be collecting blood samples to evaluate the effect that the vaccinations may have on the immune system. These tests will be done every month.
* Participants will have an MRI once every two months.
* The following tests and procedures will be done before the participant receive the vaccine and every two weeks (During the first month, these will be performed on Days 1, 3 or 4, 15, 29 and 31 or 32): medical history; physical exam; vital signs; neurological exam; routine blood tests; research blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent malignant glioma, having already been diagnosed with and treated for biopsy-proven glioblastoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed oligoastrocytoma or gliosarcoma.
* Patients will already have been treated with external beam irradiation with or without chemotherapy.
* Patients must be able to undergo a MRI.
* A priori clinical indication for open resection/debulking of recurrent malignant glioma.
* At the time of vaccination, patients must be at least 4 weeks from completion of radiotherapy and 4 weeks from cytotoxic chemotherapy.
* Serum absolute neutrophil count greater than or equal to 1500/mm3
* Serum platelets greater than or equal to 50,000/mm3
* Serum sodium greater than or equal to 125 mmol/L
* 18 years of age or older
* Karnofsky Performance Score of 60% or greater

Exclusion Criteria:

* Uncontrolled active infection
* Pregnancy or nursing mothers
* HIV infection
* Evidence of active infection with Hepatitis B or C
* Concurrent malignancy
* Active or clinically relevant autoimmune disease
* Urgent need for surgical decompression (at the time of initial consultation)
* Previous participation in a gene therapy or immunotherapy trial
* Inability to provide informed consent because of altered mental status or mental illness
* Any other medical, surgical or psychiatric condition which could interfere with the patient's inability to comply with protocol regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of preparing lethally irradiated autologous glioma cells for use in combination with irradiated GM-K562 cells as vaccination therapy in this patient population. | 3 years
To determine the safety and biological activity of subcutaneous and intradermal injection of irradiated autologous malignant glioma cells mixed with irradiated GM-CSF producing GM-K562 cells in this patient population. | 3 years

SECONDARY OUTCOMES:
Progression free survival | 3 years
overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William Curry, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts